CLINICAL TRIAL: NCT04253080
Title: Impact of the IL4I1 Enzyme Expression in Patients With Cutaneous Melanoma: Prognostic Value and/or Role in Resistance to Current Immunotherapy and Targeted Therapy
Brief Title: Expression of IL4 Induced Gene 1 in Patients With Cutaneous Melanoma: Value in Prognosis and/or in Predictive Response to Immune Checkpoint Inhibitors
Acronym: ENZYMELA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Association Robert Debré (ARD) (Unknown); Société de Dermatologie Française (Other); Institut Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP190243; 2019-A01985-52 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Cutaneous Melanoma
Keywords: cutaneous melanoma; marker for prognosis and response to targeted treatment and/or immune checkpoint inhibitor; Programmed Death ligand 1 (PD1); Cytotoxic T Lymphocyte Associated 4 (CTLA-A4)
MeSH Terms: conditions — Melanoma; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients with primary thin melanoma < or = 1mm (No Intervention): patients with primary thin melanoma (Breslow thickness less than or equal 1 mm)
- patients with primary thick melanoma > or = 3 mm (No Intervention): patients with primary thick melanoma (Breslow greater than or equal 3 mm)
- patient with melanoma who received treatment (Other): patient with melanoma (stages III or IV inoperable) and who received first line treatment with immunotherapy and / or targeted therapies
  Interventions: Biological: Blood sample; Biological: Cutaneous melanoma biopsy

INTERVENTIONS:
Biological: Blood sample — Blood sample before treatment, 3 months after treatment and after 1 year or relapse or resumption of disease progression.
  Arms: patient with melanoma who received treatment
Biological: Cutaneous melanoma biopsy — Cutaneous melanoma biopsy before treatment, 3 months after treatment and relapse or resumption of disease progression.
  Arms: patient with melanoma who received treatment

SUMMARY:
To characterize and quantify immune cells expressing the Interleukine 4 induced gene 1 (IL4I1) immunosuppressive enzyme in the blood and in tissue of melanoma patients (primary tumor, sentinel lymph nodes and cutaneous metastases).

Then, to compare the results obtained in different clinical settings:

* in cases of progression of the disease slower or faster compared to the prognosis established by clinical and pathological data
* before and after treatments with immunotherapy (anti Programmed Death ligand 1 (anti-PD1) or anti-PD1 and anti Cytotoxic T Lymphocyte associated protein 4 (anti-CTLA-4)) and / or targeted therapies (BRAF inhibitors and /or methyl ethyl ketone (MEK)).

DETAILED DESCRIPTION:
The incidence of cutaneous melanoma is increasing, but the current prognostic parameters mainly based on histological data are insufficient to identify patients with high risk of recidive. In addition, current immunotherapies using PD-1 and/or CTLA-4 antibodies have long-lasting tumor control in a substantial fraction of patients but identify new markers of treatment resistance need further investigations. Clinical data highlight enzymes involved in amino acid catabolism as new potential prognostic markers in human melanoma. Among those, the IL4I1 phenylalanine oxidase may be a new relevant marker and may represent an easily targetable molecule for cancer immunotherapy.

The current retrospective study is designed to evaluate whether a high proportion of IL4I1 positive cells within the primary tumor and/or sentinel lymph nodes allows to predict the risk of cancer recurrence from the clinical diagnosis. Immunofluorescence and immunohistochemistry will be performed.

The longitudinal study of IL4I1 positive cells in the blood and cutaneous metastasis od patients will start before and after (three months and 1 year (or before in case of treatment resistance) the treatment with targeted therapy and/or immunotherapy as a first line. Treatment will be administered on an outpatient basis. No investigational or commercial cancer directed agents or therapies other than those described below may be administered.

It is designed to evaluate whether patients that resist to treatments exhibit a high proportion of IL4I1 positive cells and how is regulated the enzyme in the course of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* group 1: patients with primary thin melanoma (Breslow thickness less than or equal to1 mm) monitored for 10 years, having relapsed or not within 10 years after the diagnosis.

  * patients with no other concomitant cancers requiring systemic treatment at the time of diagnosis of primary melanoma
  * patient or patient's family (in case of death) informed of the objectives and modalities of the study and not opposed to participation in the study
  * patient or patient's family (in case of death) not opposed to the use of part of the skin sample previously taken for the present research
* group 2: patients with primary thick melanoma (Breslow greater than or equal to 3 mm) monitored for 5 years, having relapsed or not within 5 years after diagnosis.

  * patient with no other concomitant cancers requiring systemic treatment at the time of diagnosis of primary melanoma
  * patient or patient's family (in case of death) informed of the objectives and modalities of the study and not opposed to participation in the study
  * patient or patient's family (in case of death) not opposed to the use of part of the skin sample previously taken for the present research
* group 3: patient with melanoma (stages III or IV inoperable) and who are treated with immunotherapy and / or biotherapy

  * patient with no other concomitant cancers requiring systemic treatment at the time of diagnosis of primary melanoma and initiation of systemic treatment for melanoma
  * patient informed of the objectives and modalities of the study and having given informed and written consent to participate in the study

Exclusion Criteria:

* groups 1 and 2: patient or family of the patient opposed (e) that part of the primary melanoma taken previously is used in the context of the present project
* group 3 :

  * refusal of the patient to participate in the study
  * patient unable to understand the study and sign consent
  * patient with a known contraindication to xylocaine
  * patient not affiliated to a social security system (beneficiary or beneficiary's right)
  * adult subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Role of IL4I1+ cells in prognosis and in response to treatments (targeted and/or antiPD1/CTLA4 based therapies) in cutaneous melanoma | 12 months or between 6 and 12 months (if disease progression)
  Detection of IL4I1+ cells in tissue and/or blood

CONTACTS AND LOCATIONS:
Overall Officials: Armelle Blondel, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Dermatology department, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No
The clinical data at the diagnosis and the relapse/no relapse information have to be shared from the groups 1 and 2.
  The clinical response to treatments will be shared.

REFERENCES:
- [Background] Ramspott JP, Bekkat F, Bod L, Favier M, Terris B, Salomon A, Djerroudi L, Zaenker KS, Richard Y, Molinier-Frenkel V, Castellano F, Avril MF, Prevost-Blondel A. Emerging Role of IL-4-Induced Gene 1 as a Prognostic Biomarker Affecting the Local T-Cell Response in Human Cutaneous Melanoma. J Invest Dermatol. 2018 Dec;138(12):2625-2634. doi: 10.1016/j.jid.2018.06.178. Epub 2018 Jul 23. PMID 30048651
- [Background] Bod L, Lengagne R, Wrobel L, Ramspott JP, Kato M, Avril MF, Castellano F, Molinier-Frenkel V, Prevost-Blondel A. IL4-induced gene 1 promotes tumor growth by shaping the immune microenvironment in melanoma. Oncoimmunology. 2017 Jan 13;6(3):e1278331. doi: 10.1080/2162402X.2016.1278331. eCollection 2017. PMID 28405502